CLINICAL TRIAL: NCT06265116
Title: One-Step Universal Adhesives: A 3-year Randomized Comparative Clinical Trial in Class II Composite Restorations
Brief Title: One-Step Universal Adhesives: A 3-year Clinical Trial in Class II Composite Restorations
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Omar Abd El-fattah, Phd researcher, Mansoura University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: A0801024 CD
Record Dates: First submitted 2024-02-06; First posted 2024-02-20 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-05

CONDITIONS: Dental Caries Class II; Marginal Integrity of Composite Restorations With Universal Adhesives

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Bis-GMA-containing, HEMA-containing, one-step universal adhesive. (Active Comparator): Each patient will randomly receive one class II restoration with one of the tested restorative systems
  Interventions: Other: One-step universal adhesive
- Bis-GMA-free, HEMA-containing, one-step universal adhesive (Active Comparator): Each patient will randomly receive one class II restoration with one of the tested restorative systems
  Interventions: Other: One-step universal adhesive
- Bis-GMA- free, HEMA-free, acrylic-based one-step universal adhesive (Active Comparator): Each patient will randomly receive one class II restoration with one of the tested restorative systems
  Interventions: Other: One-step universal adhesive
- Bis-GMA- containing, HEMA-containing, amide-based one-step universal adhesive (Active Comparator): Each patient will randomly receive one class II restoration with one of the tested restorative systems
  Interventions: Other: One-step universal adhesive

INTERVENTIONS:
Other: One-step universal adhesive — Each patient will receive a class II restoration using the corresponding group adhesive

SUMMARY:
to evaluate and compare the clinical performance and periodontal responses of four commercially available one-step universal adhesives with different formulations in Class II composite restorations over a three-year period.

DETAILED DESCRIPTION:
The experimental design description adhered to the guidelines provided by the Consolidated Standards of Reporting Trials (CONSORT) statement. The present study is planned as a double-blinded randomized clinical trial, ensuring that both the patients and the examiner are unaware of the treatment allocation. The trial will follow a split-mouth design. A total of forty-eight adult patients, who are seeking dental treatment, will be enrolled in the study. The participants will be recruited from the Outpatient clinic at Faculty of Dentistry, Mansoura University.

No active advertisement will be used for participant recruitment, and instead, a convenience sample will be formed. Prior to participating in the study, each patient will be required to provide informed consent by signing a consent form. The protocol of the study was approved by Mansoura University's ethics committee before initiation

ELIGIBILITY:
Inclusion Criteria:

* Patients must present with at least four posterior primary compound proximal caries involving two surfaces, specifically occluso-mesial or occluso-distal cavities, with a corresponding International Caries Detection and Assessment System (ICDAS) score of 4 or 5.
* The buccolingual width of the lesion should be approximately less than two-thirds of the intercuspal distance.
* Teeth to be restored must be in normal occlusion with the natural antagonist teeth.
* Vital teeth with no signs of pulpal inflammation or pathological lesions.
* Normal periodontal status and good oral hygiene.
* Good likelihood of recall availability.

Exclusion Criteria:

* Patients with proximal cavities that extend beyond two surfaces or have a lesion buccolingual width greater than two-thirds of the intercuspal distance, or requiring cusp coverage.
* Partly erupted or endodontic treated teeth.
* Poor oral hygiene or severe periodontitis.
* Absence of neighboring or antagonist teeth.
* Patients with known allergy to any component of the study materials.
* Patients with unstable medical conditions.
* Patients with known unavailability to attend recall visits.
* Pregnant or lactating females.
* Patients with heavy para-functional habits, fractured, or visibly cracked teeth.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2024-01-23 (Actual); Primary Completion 2027-01-23 (Estimated); Study Completion 2027-01-30 (Estimated)

PRIMARY OUTCOMES:
Percentage of functional and biological properties for each group | 3 years
  Percentage of functional and biological properties that will be clinically assessed using recently revised World Dental Federation parameters for each restorative system group

CONTACTS AND LOCATIONS:
Locations (1):
- Omar Abd El-Fattah Abd El-Maksoud, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No